CLINICAL TRIAL: NCT02845271
Title: A Two Part Protocol Using Double Blind Placebo Control to Assess the Safety, Tolerability, and Pharmacokinetics of Single Escalating Intra-articular Doses Followed by Assessment of Efficacy, Safety, Tolerability and Pharmacokinetics of a Single Intra-articular Dose of the TrkA Inhibitor, GZ389988, in Patients With Painful Osteoarthritis of the Knee
Brief Title: Proof-of-concept Study to Assess the Efficacy, Tolerability and Safety of a Single Intraarticular Dose of GZ389988 Versus Placebo in Patients With Painful Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT13830; 2014-004805-34 (EudraCT Number); U1111-1163-0806 (Other: UTN)
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Acetaminophen; Codeine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GZ389988 (Experimental): Single intraarticular injection of GZ389988 in the knee joint
  Interventions: Drug: GZ389988; Drug: acetaminophen or paracetamol; Drug: fixed combination of paracetamol + codeine; Drug: fixed combination of paracetamol + tramadol hydrochloride
- Placebo (Placebo Comparator): Single intraarticular injection of placebo for GZ389988 in the knee joint
  Interventions: Drug: placebo; Drug: acetaminophen or paracetamol; Drug: fixed combination of paracetamol + codeine; Drug: fixed combination of paracetamol + tramadol hydrochloride

INTERVENTIONS:
Drug: placebo — Pharmaceutical form:solvent for parenteral use
  Route of administration: intraarticular
  Arms: Placebo
Drug: GZ389988 — Pharmaceutical form:suspension for injection
  Route of administration: intraarticular
  Arms: GZ389988
Drug: acetaminophen or paracetamol — Pharmaceutical form: tablet
  Route of administration: oral
Drug: fixed combination of paracetamol + codeine — Pharmaceutical form: capsule
  Route of administration: oral
Drug: fixed combination of paracetamol + tramadol hydrochloride — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the efficacy of a single intraarticular dose of GZ389988 compared to placebo for relief of knee pain in patients with osteoarthritis (OA) of the knee.

Secondary Objectives:

To assess the safety and tolerability of a single intraarticular dose of GZ389988 in patients with painful OA of the knee.

To assess the pharmacokinetic parameters of a single intraarticular dose of GZ389988 in patients with painful OA of the knee.

DETAILED DESCRIPTION:
Screening will be performed within 21 days of dosing. Following the single dose of study medication, the study period for each patient will be 84 ± 7 days up to the end-of-study visit.

Total duration for one patient will be up to 16 weeks (up to the end-of-study visit), not including the long-term observational safety follow-up phone call for 12 additional weeks.

The collection of primary endpoint data up to Week 4 for futility analysis is optional. Assuming a possible step-down in dose due to safety/tolerability reasons, the total expected maximum number of included patients could be increased up to a maximum of 182 patients.

ELIGIBILITY:
Inclusion criteria :

* Men or women 40 to 80 years of age.
* Diagnosis of primary knee osteoarthritis (OA), based upon the following:
* Fulfilling the American College of Rheumatology Clinical and Radiographic criteria for OA (at least knee pain and osteophytes), with
* X-ray evidence within the last 6 months for Kellgren and Lawrence classification II to IV.
* Western Ontario and McMaster Universities Arthritis Index (WOMAC) A1 Pain subscore (walking pain) over the last 48 hours ≥40 and ≤90 on VAS 0-100 in the target knee at screening with or without medication, and ≤30 on Visual Analogue Scale (VAS) 0-100 in the contralateral knee at screening with or without medication.
* WOMAC A1 pain subscore (walking pain) between 50 and 90 using the VAS 0-100, corresponding to moderate to severe pain in the target knee at baseline (from eDiary, average of at least 3 days in the time window between Day-5 and Day-1).
* Symptomatic for more than 6 months (if both symptomatic knees, at least for the most painful knee that will receive the study drug).
* Having given written informed consent prior to any procedure related to the study.
* Ambulatory with an active lifestyle and in good general health. (Assistive devices were allowed if used throughout a period of 3 months or more prior to screening, on the condition that they continue to be used throughout the study).
* A male who is sexually active must use a condom as part of a method of highly effective contraception (eg, condom + spermicide, and an additional contraceptive method used by the partner) during sexual intercourse with a women of childbearing potential for the duration of the study period up to the end-of-study visit and should not father a child in this period. Male patients also have to agree not to donate sperm for the duration of the study until the end-of-study visit.

Exclusion criteria:

* Women of childbearing potential.
* Pregnant or breastfeeding women.
* Any uncontrolled, chronic condition or laboratory finding which, in the opinion of the Investigator, could potentially put the patient at increased risk.
* Patients with clinically significant or uncontrolled hepatic, gastrointestinal, cardiovascular, respiratory, neurological (including diabetic neuropathy), psychiatric, hematological, renal, or dermatological disease, or any other medical condition, such as symptomatic peripheral vascular disease of the study leg (prior or current), clinically significant venous or lymphatic stasis present in the study leg, that might interfere with the evaluation of investigational medicinal product (IMP) according to Investigator's medical judgment.
* Chondrocalcinosis.
* Fibromyalgia.
* Moderately severe or severe depression as indicated by Patient Health Questionnaire-9 (PHQ-9) total score at screening visit.
* Severe anxiety as indicated by Generalized Anxiety Disorder (GAD-7) score at screening visit.
* History or presence of drug or alcohol abuse (alcohol consumption >40 grams per day).
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development, or unable to use an electronic diary daily.
* Abnormal coagulation parameters: outside the range international normalized ratio (INR) 0.85-1.15, activated partial thromboplastin time >33 seconds, platelets <140 x 10^9/L.
* Moderate to severe renal impairment.
* Underlying hepatobiliary disease and/or alanine aminotransferase (ALT) >2 x upper limit of normal (ULN).
* High sensitivity C-reactive protein (hsCRP) >2 x ULN.
* Hemoglobin <10 g/dL, white blood cell count (WBC) <3 x 10^9/L.
* Positive result on any of the following tests: hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Secondary OA. -Ipsilateral hip OA.-
* History of osteonecrosis and/or rapidly progressive OA (RPOA).
* Intraarticular injection within 3 months prior to inclusion.
* Unable to be maintained for at least 2 weeks prior to entry into study on paracetamol (no non-steroidal anti-inflammatory drug [NSAID] use during the 12 weeks of the study; after the end-of-study visit [Day 84 ± 7] patients may be given an NSAID if necessary to provide better control of OA symptoms).
* Any IMP within 3 months prior to the study.
* Any knee magnetic resonance imaging (MRI) contraindication.
* Patients at risk of developing a RPOA with pre-existing findings on MRI of the target knee at baseline.
* Patients with pain DETECT questionnaire (PD-Q) score >18.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly mean score of Western Ontario and McMaster Universities Arthritis Index (WOMAC) A1 pain subscore (walking pain) collected daily in the target knee, as measured by the Visual Analogue Scale (VAS) 0-100 | Averaged over 4 weeks (up to Day 28)

SECONDARY OUTCOMES:
Change from baseline in weekly mean score of WOMAC A1 pain sub-score (walking pain) collected daily in the target knee, as measured by the VAS 0-100 | Averaged over 12 weeks (up to Day 84)
Change from baseline in weekly mean score of WOMAC A1 pain sub-score collected daily in the target knee | Averaged over 1, 2, 3, 6, 8, and 10 weeks
Change from baseline in weekly mean score of WOMAC A1 pain sub-score collected daily in the target knee | At 1, 2, 3, 4, 6, 8, 10, and 12 weeks
Change from baseline in weekly mean score of overall knee pain collected daily in the target knee | At and averaged over 1, 2, 3, 4, 6, 8, 10, and 12 weeks
Change from baseline in Patient Global Assessment (PGA) of disease status | At and averaged over 1, 2, 3, 4, 6, 8, 10, and 12 weeks
Change from baseline in WOMAC index (total score for pain, stiffness, and physical function subscales), pain, stiffness and physical function sub-scores | Averaged over 1, 2, 3, 4, 6, 8, 10, and 12 weeks
Patient Global Impression of Change (PGIC) | Over the last 4 weeks at Day 28 (1 to 4 weeks), Day 56 (5 to 8 weeks), and Day 84 (9 to 12 weeks)
Patient Global Assessment of Response to Therapy (PGART) | Over the last 4 weeks at Day 28 (1 to 4 weeks), Day 56 (5 to 8 weeks), and Day 84 (9 to 12 weeks)
Rate of response to therapy according to Outcome Measures in Rheumatology committee (OMERACT) and the Osteoarthritis Research Society International (OARSI) | By Day 28, Day 56, and Day 84
  OMERACT and OARSI responder criteria are based on the symptomatic variables pain and function, or pain, function and patient's global assessment
WOMAC A1 responder rate based on percentage of patients with reduction in pain intensity of at least 30% and 50% at endpoint compared to baseline | Over 4 weeks (up to Day 28) and 12 weeks (up to Day 84) and at 1, 2, 3, 4, 6, 8, 10, and 12 weeks
Time to first WOMAC A1 response for ≥30% reduction in pain intensity | At 1, 2, 3, 4, 6, 8, 10, 12 weeks
Time to first WOMAC A1 response for 50% reduction in pain intensity | At 1, 2, 3, 4, 6, 8, 10, 12 weeks
Amount of rescue medication intake | Up to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Germany (2):
  - Investigational Site Number 276001, Berlin
  - Investigational Site Number 276002, Lübeck

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Krupka E, Jiang GL, Jan C. Efficacy and safety of intra-articular injection of tropomyosin receptor kinase A inhibitor in painful knee osteoarthritis: a randomized, double-blind and placebo-controlled study. Osteoarthritis Cartilage. 2019 Nov;27(11):1599-1607. doi: 10.1016/j.joca.2019.05.028. Epub 2019 Jul 25. PMID 31351965